CLINICAL TRIAL: NCT04430257
Title: Efficacy of a Community-based PrEP Uptake Intervention for People Who Inject Drugs (PWID) in the US Northeast
Brief Title: Pre-exposure Prophylaxis (PrEP) for Health
Acronym: PrEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Fenway Institute (Other); AIDS Action Committee of Massachusetts (Other); Greater Lawrence Family Health Center (Unknown); University of California, San Diego (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011002841; R01DA051849-01 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Substance Dependence; HIV (Human Immunodeficiency Virus)
Keywords: PrEP (pre-exposure prophylaxis ); PWID (people who inject drugs); SSP (syringe service program); HIV education; Motivational interviewing; Self efficacy; Social cognitive theory
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — Seroconversion; Motivational Interviewing; Patient Navigation; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals collecting the primary outcome data will be blinded to intervention condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrEP for health (Experimental): Participants in the PrEP (pre-exposure prophylaxis) for health arm will receive theory informed HIV and PrEP education, motivational interviewing, problem-solving and planning, and ongoing patient navigation.
  Interventions: Other: HIV and PrEP education; Behavioral: Motivational interviewing; Behavioral: Problem-solving and planning; Behavioral: Patient navigation; Other: PrEP information
- Standard of care (Active Comparator): Participants in the standard of care arm will receive PrEP information and referrals.
  Interventions: Other: PrEP information; Other: Referrals

INTERVENTIONS:
Other: HIV and PrEP education — Navigators will deliver Social Cognitive Theory-informed HIV and PrEP education.
  Arms: PrEP for health
Behavioral: Motivational interviewing — Bachelors-level PrEP Navigators who are trained in motivational interviewing (MI) will use MI to promote the behavioral intervention.
  Arms: PrEP for health
Behavioral: Problem-solving and planning — Bachelors-level PrEP Navigators will assist participants with problem-solving and planning.
  Arms: PrEP for health
Behavioral: Patient navigation — Ongoing PrEP navigation support to promote participants' initial and continued engagement with PrEP clinics affiliated with the two study sites
  Arms: PrEP for health
Other: PrEP information — A brief video that describes what PrEP is and how it works to prevent HIV via sexual and injection transmission will be shown to participants.
Other: Referrals — Study staff will provide basic information about PrEP and referrals to PrEP clinicians.
  Arms: Standard of care

SUMMARY:
This randomized controlled trial will test the efficacy of "PrEP for Health," a behavioral intervention to improve the use of antiretroviral pre-exposure prophylaxis (PrEP) among at-risk people who inject drugs (PWID) in two syringe service program (SSP) settings in Lawrence and Boston/Cambridge, Massachusetts. The investigators will equally randomize 200 PWID to receive either (a) the "PrEP for Health" intervention condition involving theory-informed HIV and PrEP education, motivational interviewing, problem-solving and planning, and ongoing patient navigation (n=100), or (b) the standard of care condition involving PrEP information and referrals (n=100). Successful PrEP uptake (via medical/pharmacy records), post-treatment PrEP adherence (assessed at 3 months via drug levels in hair), and longer-term PrEP adherence (assessed at 6 and 12 months via drug levels in hair) will be evaluated. The degree to which intervention efficacy occurs through specific conceptual mediators and differs according to hypothesized moderators will also be evaluated.

DETAILED DESCRIPTION:
The overall goal of this proposal is to evaluate the efficacy of the "PrEP for Health" navigator delivered behavioral intervention in improving PrEP uptake (via medical/pharmacy records), post-treatment PrEP adherence (assessed at 3 months via drug levels in hair), and longer-term PrEP adherence (assessed at 6 and 12 months via drug levels in hair) among PWID in SSPs. Eligible PWID (n=200 total; 100 recruited from each study site) will be equally randomized to an active PrEP for Health intervention arm (n=100) or a Standard of Care control condition (n=100). Assessments will be conducted at baseline and 1, 3, 6, and 12 months after randomization.

We hypothesize that brief, multi-component behavioral intervention sessions with ongoing support delivered by trained PrEP Navigators within Syringe Service Programs (SSPs) will improve PrEP uptake, adherence, and long-term adherence in PWID by increasing HIV and PrEP knowledge (including alleviating concerns about side effects), increasing HIV risk perceptions and PrEP interest and motivation, improving PrEP use self-efficacy and behavioral skills, and reducing structural barriers over time. Based on our formative research, we also hypothesize that the strength of intervention effects may differ by key individual characteristics (age, gender, baseline sexual risk, polysubstance, and stimulant use).

This is a randomized control trial (RCT). Participants will be recruited via outreach specialist at SSP sites and during routine community outreach practices of the organizations. After eligibility confirmation and baseline assessments, participants will be randomized to one of two study arms: 1) Standard of Care (SOC) Control Condition: as routinely provided through the SSP study sites, participants will receive information and services according to routine practice and a brief video that describes what PrEP is and how it works to prevent HIV via sexual and injection transmission; 2) "PrEP for Health" Intervention Condition: a trained PrEP Navigator will deliver a manualized PrEP uptake and adherence intervention in private counseling rooms at SSPs followed by 3 months of additional PrEP navigation support through in-person, phone, and text interactions as needed. Participants will complete a total of four follow-up visits over a 12-month period. Participants who initiate PrEP will have a hair sample collected at 3-, 6-, and 12-month visits. All participants will receive a rapid HIV screening test at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected (verified by rapid/4th generation test)
* Reporting past-month injection of any drugs
* One or more HIV risk behaviors (past-month receptive syringe sharing, transactional sex, or condomless sex with an HIV-infected or unknown-status partner)
* Not currently on and never taken PrEP
* Able to understand and speak English or Spanish

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness, cognitive impairment, or substance intoxication at the time of enrollment
* Living in Massachusetts (MA) for <3 months
* Planning to move out of MA within a year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | 3 months
  PrEP uptake will be assessed via medical/pharmacy records
Post-treatment PrEP adherence | 3 months
  PrEP adherence will be assessed by drug levels in hair samples at the acute follow up time point (3 months post-baseline)

SECONDARY OUTCOMES:
Longer-term PrEP adherence | 6 and 12 months
  Longer-term PrEP adherence will be assessed by drug levels in hair samples at 6 and 12-month post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katie Biello, PhD, MPH, Principal Investigator — Brown University; Angela Bazzi, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - AIDS Action, Cambridge, Massachusetts
  - Greater Lawrence Family Health Center, Lawrence, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
By request to the study investigators
Time Frame: Data will be available after the study has closed and after publication of the primary study findings.
Access Criteria: Requests will be reviewed by the principal investigators.

REFERENCES:
- [Derived] Bazzi AR, Bordeu M, Baumgartner K, Sproesser DM, Bositis CM, Krakower DS, Mimiaga MJ, Biello KB. Study protocol for an efficacy trial of the "PrEP for Health" intervention to increase HIV PrEP use among people who inject drugs. BMC Public Health. 2023 Mar 17;23(1):513. doi: 10.1186/s12889-023-15429-w. PMID 36932369